CLINICAL TRIAL: NCT07182539
Title: Atelectasis in Pediatric Anesthesia: A Randomized Observational Study Comparing Volume-Controlled and Pressure-Regulated Volume Control Ventilation Via Lung Ultrasound and Electrical Impedance Tomography
Brief Title: VCV vs PRVC in Pediatric Anesthesia; an EIT- and LS-based Study
Acronym: VentiEIT_ped
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vittore Buzzi Children's Hospital (Other)
Responsible Party: Principal Investigator, Anna Camporesi, Medical Coordinator of Pediatric Anesthesia, Vittore Buzzi Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: VentiEIT_ped
Record Dates: First submitted 2025-08-02; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Atelectasis
Keywords: Atelectasis; Lung Ultrasound; EIT; Pediatric Anesthesia
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Randomization: Eligible patients will be randomized in an equal manner (1:1) to receive Volume Control Ventilation (VCV) or Pressure Regulated Volume Control (PRVC/PCV-VG). The randomization sequence will be generated by a computerized system to ensure unpredictability of the assignment. Randomization will be managed by an independent investigator not involved in direct patient care or data collection and will be stratified by center.
Who Masked: Participant
Masking Description: Patients will not be aware of the randomization arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRVC ventilation (Experimental): Patients in this arm will be ventilated in PRVC.
  Interventions: Other: PRVC ventilation
- VCV ventilation (Active Comparator): Patients in this arm will be ventilated in VCV.
  Interventions: Other: VCV ventilation

INTERVENTIONS:
Other: PRVC ventilation — Ventilation in PRVC mode.
  Arms: PRVC ventilation
Other: VCV ventilation — Ventilation in VCV mode.
  Arms: VCV ventilation

SUMMARY:
The primary objective of this study is to evaluate and compare the incidence and severity of intraoperative pulmonary atelectasis, measured by Lung Ultrasound Score (LUS) and EIT (Electrical Impedance Tomography), between two different modes of mechanical ventilation: Volume Control Ventilation (VCV) and Pressure Regulated Volume Control (PRVC/PCV-VG)

DETAILED DESCRIPTION:
Background Mechanical ventilation is often required in pediatric anesthesia. However, the optimal intraoperative ventilatory strategy for pediatric patients remains a matter of debate, with no definitive consensus to date. Among conventional modes, Pressure-Controlled Ventilation (PCV) is time-triggered, pressure-limited, time cycled; set parameters include peak inspiratory pressure (PIP), inspiratory time (Ti) and respiratory rate (RR). Tidal Volume (TV) is a dependent variable. With the constant pressure throughout inspiration, PCV is thought to provide the maximum inspiratory pressure for the entire inspiratory-time favoring lung recruitment1.

In contrast, Volume-Controlled ventilation (VCV) delivers the preset TV, and the PIP is dependent on the respiratory mechanics of the patient. VCV has the advantage of certain TV delivery, while PCV has the advantage of not exceeding the set PIP1.

Both have limitations and to overcome the inherent compromises of traditional modes, modern ventilation modes such as Pressure Regulated Volume Control (PRVC) have been developed. These modes are designed to combine the benefits of VCV and PCV. They use a pressure-controlled flow and ventilation application approach, integrated with digital feedback mechanisms that continuously monitor the applied tidal volume, targeting a fixed tidal volume. PRVC allows the ventilator to measure the patient's lung compliance on a breath-to-breath basis and determine the pressure required to be given for the set Ti to achieve the set tidal volume. As a result, the ventilator can deliver a square wave pressure waveform like PCV but also ensure that a constant tidal volume is delivered to the patient like VCV.

Regardless of the ventilation strategy, general anesthesia inevitably induces atelectasis2, due to different mechanisms such as: shift of the diaphragm towards the thorax thus causing compressions of some lung areas, surfactant alteration due to inhalational anaesthetics, high inspired fractions of oxygen (FiO2) which are reabsorbed from the alveoli into the bloodstream causing reduction of the alveolar size3. These effects are demonstrable both immediately after induction and at the endo of surgery.

Children are particularly vulnerable to anaesthesia-induced atelectasis, due to the relatively higher compliant chest wall and the presence of diaphragmatic compression by large abdominal organs4. The clinical consequences of atelectasis are significant and include increased intrapulmonary shunt (blood passing through the lungs without being oxygenated), perioperative desaturation, higher risk of pneumonia, and a broader spectrum of postoperative pulmonary complications (PPCs)5. Given the peculiarities that predispose paediatric patients to atelectasis, they cannot be considered simply as miniature adults; their unique physiology requires tailored protective ventilation strategies. This highlights the urgency of identifying optimal ventilatory modes capable of minimizing atelectasis in this vulnerable population Since the best ventilatory strategy to avoid atelectasis is not defined currently, with the present randomized clinical trial the investigators aim to compare the effects of two ventilatory modes (VCV and PRVC) at same settings in terms of tidal volume, PEEP, FiO2, on atelectasis as described by lung ultrasound and EIT. The investigators hypnotized that PRVC (combining pressure control with guaranteed tidal volume) reduces atelectasis severity compared to VCV, as measured by LUS and EIT.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring intraoperative mechanical ventilation via endotracheal intubation
* Written informed consent obtained from parents or legal guardians. For children capable of understanding, assent will also be obtained based on age and cognitive ability.
* ASA (American Society of Anesthesiologists) physical status I-II

Exclusion Criteria:

* Patients with significant pre-existing lung disease (e.g., cystic fibrosis, severe bronchopulmonary dysplasia, severe uncontrolled asthma, neuromuscular disease with respiratory compromise).
* Patients with complex congenital heart disease or significant hemodynamic instability.
* Patients undergoing thoracic surgery or procedures that could significantly alter lung mechanics (e.g., pre-existing pneumothorax).
* Refusal of parents/guardians or patient to participate in the study.
* History of previous intrathoracic procedure.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Atelectasis at lung ultrasound | From baseline to recovery in post-anesthesia care unit
  To compare the incidence of intraoperative pulmonary atelectasis, measured by Lung Ultrasound Score (LUS) , between two different modes of mechanical ventilation: Volume Control Ventilation (VCV) and Pressure Regulated Volume Control (PRVC/PCV-VG).
Atelectasis | From baseline to recovery in post-anesthesia care unit
  To compare the severity of intraoperative pulmonary atelectasis, measured by EIT, between two different modes of mechanical ventilation: Volume Control Ventilation (VCV) and Pressure Regulated Volume Control (PRVC/PCV-VG).

SECONDARY OUTCOMES:
Regional distribution of ventilation and lung homogeneity | From baseline to recovery in post-anesthesia care unit
  Compare regional distribution of ventilation between VCV and PRVC groups. This will be accomplished using parameters derived from Thoracic Electrical Impedance (EIT), such as Global Inhomogeneity Index (GI) and center of ventilation (CoV).
Peak Inspiratory Pressure | From baseline to recovery in post-anesthesia care unit
  Evaluate the impact of the two ventilation modes on Peak Inspiratory Pressure (PIP).
Plateau Pressure | From baseline to recovery in post-anesthesia care unit
  Evaluate the impact of the two ventilation modes on Plateau Pressure.
Static Respiratory System Compliance | From baseline to recovery in post-anesthesia care unit
  Evaluate the impact of the two ventilation modes on Static respiratory System Compliance
Dynamic Respiratory System Compliance | From baseline to recovery in post-anesthesia care unit
  Evaluate the impact of the two ventilation modes on Dynamic respiratory System Compliance

CONTACTS AND LOCATIONS:
Locations (1):
- Vittore Buzzi Children's Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Camporesi A, Roveri G, Vetrugno L, Buonsenso D, De Giorgis V, Costanzo S, Pierucci UM, Pelizzo G. Lung ultrasound assessment of atelectasis following different anesthesia induction techniques in pediatric patients: a propensity score-matched, observational study. J Anesth Analg Crit Care. 2024 Oct 5;4(1):69. doi: 10.1186/s44158-024-00206-x. PMID 39369249
- [Background] Frerichs I, Schiffmann H, Hahn G, Hellige G. Non-invasive radiation-free monitoring of regional lung ventilation in critically ill infants. Intensive Care Med. 2001 Aug;27(8):1385-94. doi: 10.1007/s001340101021. PMID 11511953
- [Background] Kim YS, Won YJ, Lee DK, Lim BG, Kim H, Lee IO, Yun JH, Kong MH. Lung ultrasound score-based perioperative assessment of pressure-controlled ventilation-volume guaranteed or volume-controlled ventilation in geriatrics: a prospective randomized controlled trial. Clin Interv Aging. 2019 Jul 18;14:1319-1329. doi: 10.2147/CIA.S212334. eCollection 2019. PMID 31409981
- [Background] Bauer M, Opitz A, Filser J, Jansen H, Meffert RH, Germer CT, Roewer N, Muellenbach RM, Kredel M. Perioperative redistribution of regional ventilation and pulmonary function: a prospective observational study in two cohorts of patients at risk for postoperative pulmonary complications. BMC Anesthesiol. 2019 Jul 27;19(1):132. doi: 10.1186/s12871-019-0805-8. PMID 31351452